CLINICAL TRIAL: NCT06167863
Title: Retrospective Analysis of the Correlation Between CT/MRI Imaging Features and Pathology, Prognosis in Patients With Renal Tumors
Brief Title: Retrospective Analysis of the Correlation Between Imaging Features and Pathology, Prognosis in Renal Tumors
Status: Completed | Type: Observational
Sponsor: Zhen Li (Other)
Responsible Party: Sponsor-Investigator, Zhen Li, professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20230893
Record Dates: First submitted 2023-11-30; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Radiomics; Deep Learning; Artificial Intelligence; Body Composition
MeSH Terms: interventions — Radiomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WHO ISUP grading high: high-grade refer to Grades 3 and 4 tumours with an unfavourable prognosis
  Interventions: Diagnostic Test: radiomics
- WHO ISUP grading low: low-grade refer to Grades 1 and 2 tumours with a promising prognosis
  Interventions: Diagnostic Test: radiomics

INTERVENTIONS:
Diagnostic Test: radiomics — extracted image features from CT or MRI

SUMMARY:
Renal cell carcinoma (RCC) is the most common malignant tumor in the kidney with a high mortality rate. Traditional imaging techniques are limited in capturing the internal heterogeneity of the tumor. Radiomics provides internal features of lesions for precise diagnosis, prognosis prediction, and personalized treatment planning. Early and accurate diagnosis of renal tumors is crucial, but it's challenging due to morphological and pathological overlap between benign and malignant lesions. The accurate diagnosis of RCC, especially for small tumors, remains a significant challenge. Recent studies have shown a relationship between body composition, obesity, and renal tumors. Common indicators like body weight and BMI fail to reflect body composition accurately. Research on the role of body composition, including adipose tissue, in tumor pathology could improve clinical diagnosis and treatment planning.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) accounts for 80-90% of malignant tumors in the kidney and has the highest mortality rate among genitourinary tumors. Imaging examinations play an important role in the diagnosis, preoperative assessment, selection of surgical methods, and evaluation of therapeutic efficacy in RCC. However, traditional imaging primarily reflects the morphological and functional changes of the tumor and cannot reflect the internal heterogeneity. In the current era of precision medicine, radiomics can provide internal features of lesions that cannot be observed by the naked eye, enabling precise diagnosis, prognosis prediction, efficacy evaluation, and personalized treatment planning for tumors. Renal cell carcinoma is highly elusive, with over 30% of patients already experiencing metastasis at the time of initial diagnosis, and it is insensitive to radiotherapy and chemotherapy. Early diagnosis and differential diagnosis of renal tumors are important prognostic factors that affect patient survival and treatment. Given the different treatment approaches, preoperative differentiation of lesion nature holds significant clinical significance. However, there is some overlap in the morphological and pathological features between benign and malignant lesions of the kidney, making it difficult to differentially diagnose such tumors using existing imaging techniques alone. Therefore, the accurate diagnosis of renal cell carcinoma, especially for small renal tumors (≤4cm), remains a significant challenge. In recent years, the relationship between body composition, such as obesity, and renal tumors has received increasing attention. Previous studies have shown a close association between obesity and kidney cancer. Common indicators such as body weight, BMI, and waist circumference fail to effectively reflect body composition, including various fat and muscle distributions and relative amounts. Different body compositions have different physiological functions and varying impacts on tumors. Further specific research on the true role of various body compositions, including adipose tissue, in tumor pathology would aid in clinical diagnosis and subsequent treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Our hospital admits patients with renal tumors in the urology department. The diagnosis is confirmed through surgical pathology, and the patients' imaging data is obtained through contrast-enhanced Computed Tomography or Magnetic Resonance examination in the radiology department.

Exclusion Criteria:

* Patients who have undergone puncture, microwave, interventional therapies before the examination, or who have received chemotherapy or radiotherapy;
* Patients with poor respiratory coordination, resulting in significant image artifacts;
* Lesions are cystic, without discernible regions of interest, or with multiple regions of necrosis within the lesion;
* Lesions are too small, with a diameter of less than 1cm;
* Thin-slice imaging is not available in the CT scan.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with renal tumors
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
WHO/ISUP grade pathologically | 1 month
  The WHO ISUP grade of the tumor indicated in the post-operative surgical pathology report

SECONDARY OUTCOMES:
pathological T stage | 1 month
  pathological T stage according to the eighth TNM system.

CONTACTS AND LOCATIONS:
Overall Officials: Li Dr, Principal Investigator — Tongji Hospital
Locations (1):
- Zhen Li, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li S, Zhou Z, Gao M, Liao Z, He K, Qu W, Li J, Kamel IR, Chu Q, Zhang Q, Li Z. Incremental value of automatically segmented perirenal adipose tissue for pathological grading of clear cell renal cell carcinoma: a multicenter cohort study. Int J Surg. 2024 Jul 1;110(7):4221-4230. doi: 10.1097/JS9.0000000000001358. PMID 38573065